CLINICAL TRIAL: NCT00304681
Title: The Effectiveness of CONCERTA® vs. Usual Clinical Care With Immediate Release Methylphenidate (IR MPH) in Children (6-12 Years) With Attention Deficit Hyperactivity Disorder (ADHD): A Randomized, Open-Label Trial
Brief Title: An Effectiveness and Safety Study of CONCERTA* vs. Immediate Release Methylphenidate (IR MPH) in Attention Deficit Hyperactivity Disorder Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Ortho Inc., Canada (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR003112
Record Dates: First submitted 2006-03-17; First posted 2006-03-20 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2010-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; OROS* Methylphenidate
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

INTERVENTIONS:
Drug: OROS*-Methylphenidate

SUMMARY:
The purpose of this study is to determine the effectiveness and safety of OROS*methylphenidate/CONCERTA* vs. immediate release methylphenidate as a treatment for ADHD specifically for those children who have behavioural difficulties in the afternoon/after-school and evening periods.

DETAILED DESCRIPTION:
Methylphenidate, namely immediate release methylphenidate is the primary stimulant used in the treatment of children with Attention Deficit Hyperactivity Disorder (ADHD). Immediate release methylphenidate has limitations related to its time course of action.As the morning dose wears off, inattention may increase during late-morning classes. Similarly, when the midday dose is wearing off, the child may experience difficulty concentrating on homework. The second problem relates to compliance with midday and late afternoon dosing. Children feel stigmatized or embarrassed by trips to the nurse's office for medication and may skip doses as a result. In other cases, a school nurse may not be available or policies prohibit staff from administering drugs so children may be required to self-administer drug. CONCERTA® was developed to overcome these limitations. The purpose of this study is to see how effective and safe Concerta* is vs. immediate release methylphenidate in children with ADHD.

Patients will take either Concerta* (18, 27, 36, or 54 mg) or Immediate Release Methylphenidate tablets (maximum 60mg/day) orally every morning for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be between 6 and 12 years of age inclusive, have a diagnosis of Attention Deficit Hyperactivity Disorder (ADHD) as defined by the DSM-IV established through clinical interview by the investigator and corroborated by the SNAP-IV parent rating scale, who in the opinion of the parents/caregivers exhibit significant after-school/evening behavioural difficulties where 12 hour coverage is desired
* Eligible patients will be evaluated after a minimum 3 day washout period without ADHD medication
* In addition, patients must also have a CGI-Severity score, at baseline of "moderate", "marked", "severe" or "extremely severe" in order to be eligible
* Patients could have had no prior treatment for ADHD or are presently taking something or could have had ADHD medication treatment in the past

Exclusion Criteria:

* No patients with marked anxiety, tension, aggression or agitation, glaucoma, an ongoing seizure disorder, a psychotic disorder, a diagnosis of Tourette's disorder, or a family history of Tourette's disorder, bipolar disorder, suspected mental retardation, significant learning disability, eating disorder or history of one, pre-existing gastrointestinal narrowing
* No patient with inability to swallow the medication whole, those with any unstable medical illness were excluded

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 147 (Actual)
Dates: Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Change in average SNAP-IV(Swanson, Nolan and Pelham -IV) score from baseline at end of study and the remission of symptoms between groups, defined as an average SNAP-IV score of <=1 at end of study

SECONDARY OUTCOMES:
changes at end of study for Parenting Stress Index, Conners Parent Rating Scale, IOWA Conners Parent Rating Scale, Visual Analogue Scale for homework and social play, Resource Use Questionnaire, parent satisfaction, Clinical Global Impression

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Ortho Inc. Clinical Trial, Study Director — Janssen-Ortho Inc., Canada

REFERENCES:
- [Result] Steele M, Weiss M, Swanson J, Wang J, Prinzo RS, Binder CE. A randomized, controlled effectiveness trial of OROS-methylphenidate compared to usual care with immediate-release methylphenidate in attention deficit-hyperactivity disorder. Can J Clin Pharmacol. 2006 Winter;13(1):e50-62. Epub 2006 Jan 23. PMID 16456216
- See also: A Randomized, Controlled, Effectiveness Trial of OROS-Methylphenidate compared to Usual Care with Immediate-Release-Methylphenidate in Attention-Deficit-Hyperactivity-Disorder — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=358&filename=CR003112_CSR.pdf